CLINICAL TRIAL: NCT04509466
Title: A Multicentre, Open-label, Single-arm, Phase I/II Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of Liposomal Mitoxantrone Hydrochloride Injection Combined With Pegaspargase in the Treatment of NKTCL
Brief Title: Clinical Study of Liposomal Mitoxantrone Hydrochloride Injection Combined With Pegaspargase in the Treatment of NKTCL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-012
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2020-08

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dose escalation (part 1) (Experimental): dose escalation (part 1):Patients with treatment-naïve, relapsed or refractory extranodal natural killer/T-cell lymphoma (nasal type) will receive liposomal mitoxantrone hydrochloride plus a standard dose of pegaspargase every 21 days (a cycle) for a maximum of 6 cycles. The starting dose of liposomal mitoxantrone hydrochloride is 12mg/m2.dose expansion, treatment-naïve patients (part 2):Patients with treatment-naïve extranodal natural killer/T-cell lymphoma (nasal type) will receive liposomal mitoxantrone hydrochloride at RP2D plus a standard dose of pegaspargase every 21 days (a cycle) for a maximum of 6 cycles.
  dose expansion, relapsed or refractory patients (part 2):Patients with relapsed or refractor extranodal natural killer/T-cell lymphoma (nasal type) will receive liposomal mitoxantrone hydrochloride at RP2D plus a standard dose of pegaspargase every 21 days (a cycle) for a maximum of 6 cycles.
  Interventions: Drug: Part 1: Liposomal mitoxantrone hydrochloride and Pegaspargase; Drug: Part 2 (treatment-naïve patients): Liposomal mitoxantrone hydrochloride and Pegaspargase; Drug: Part 2 (relapsed or refractory patients): Liposomal mitoxantrone hydrochloride and Pegaspargase

INTERVENTIONS:
Drug: Part 1: Liposomal mitoxantrone hydrochloride and Pegaspargase — Drug: Liposomal mitoxantrone hydrochloride (12mg/m2, 16mg/m2, 20mg/m2, 24mg/m2) is administered by an intravenous infusion (IV) on day 1 of each 21-day cycle.
  Drug: Pegaspargase (2000IU/m2) is administered by an intramuscular injection (IM) on day 1 of each 21-day cycle.
  Other Names: Part 1
Drug: Part 2 (treatment-naïve patients): Liposomal mitoxantrone hydrochloride and Pegaspargase — Drug: Liposomal mitoxantrone hydrochloride (RP2D defined in Part 1) is administered by an intravenous infusion (IV) on day 1 of each 21-day cycle.
  Drug: Pegaspargase (2000IU/m2) is administered by an intramuscular injection (IM) on day 1 of each 21-day cycle.
  Other Names: Part 2 (treatment-naïve patients)
Drug: Part 2 (relapsed or refractory patients): Liposomal mitoxantrone hydrochloride and Pegaspargase — Drug: Liposomal mitoxantrone hydrochloride (RP2D defined in Part 1) is administered by an intravenous infusion (IV) on day 1 of each 21-day cycle.
  Drug: Pegaspargase (2000IU/m2) is administered by an intramuscular injection (IM) on day 1 of each 21-day cycle.
  Other Names: Part 2 (relapsed or refractory patients)

SUMMARY:
This is a multicentre, open-label, single-arm, phase I/II clinical study to evaluate the safety, efficacy and pharmacokinetics of liposomal mitoxantrone hydrochloride in combination with pegaspargase in patients with extranodal natural killer/T-cell lymphoma, nasal type (NKTCL).

DETAILED DESCRIPTION:
This is a multicentre, open-label, single-arm, phase I/II clinical study with a dose-escalation stage (part 1) and a dose-expansion stage (part 2). In part 1, patients with treatment-naïve, relapsed/refractory extranodal natural killer/T-cell lymphoma (nasal type) will be assigned to receive sequentially higher doses of liposomal mitoxantrone hydrochloride plus a standard dose of pegaspargase every 21 days (a cycle). The dose escalation initially will follow an accelerated titration design for the first two dosing groups, then follow a classic 3+3 design. All dose-escalation decisions will be based on the safety data generated from the currently highest dose group. The maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of liposomal mitoxantrone hydrochloride will be determined in part 1. In part 2, additional patients will be recruited into two groups,the treatment-naïve group and the relapsed or refractory group, to receive liposomal mitoxantrone hydrochloride at the RP2D combined with a standard dose of pegaspargase. All patients will receive the treatment until disease progression, or observation of unacceptable grade 3 drug-related adverse events (a maximum of 6 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18, ≤75 years, no gender limitation;
3. Histologically confirmed diagnosis of treatment-naïve, relapsed or refractory extranodal NK/T-cell lymphoma nasal type (NKTCL);
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
5. At least one measurable lesion as per Lugano 2014 criteria;
6. Adequate bone marrow, liver, renal and coagulation function

Exclusion Criteria:

1. Known central nervous system involvement caused by lymphoma;
2. Known infiltration of the bone marrow according to criteria for leukemia (≥20% myeloblast in the blood or bone marrow);
3. Known hemophagocytic syndrome;
4. History of allergy and contraindications to mitoxantrone hydrochloride and/or asparaginase/ pegaspargase;
5. Chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatment within 4 weeks of the first dose of the study drug (2 weeks for the local radiation therapy for pain relief);
6. Life expectancy < 3 months
7. Impaired cardiac function or serious cardiac disease;
8. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or other active viral infection;
9. Acute symptomatic or chronic pancreatitis within 4 weeks prior to screening;
10. History of, or known additional tumor (exception: non-melanoma skin cancer (in situ) and cervical cancer (in situ) which have been cured and have not recurred within 5 years);
11. History of solid organ transplantation, autologous hematopoietic stem cell transplantation within 6 months prior to screening, or allogeneic hematopoietic stem cell transplantation before screening;
12. Major surgery within 4 weeks prior to screening. Or have a surgical schedule during the study period;
13. A serious infection within 4 weeks prior to screening and not suitable for the study according to the judgment of the investigator;
14. Uncontrolled diabetes at screening;
15. Known alcohol or drug abuse;
16. Known psychiatric disorders or cognitive disorder;
17. 17. Pregnant or breastfeeding women, or patients who are expecting to conceive or father in 12 months (starting with the screening visit)；
18. Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Part 1：dose limiting toxicities (DLTs) | Cycle 1 (a cycle = 21 days)
  The incidence and severity of adverse events (AEs), abnormalities in clinical laboratory assessments, ECGs, vital sign assessments, and physical exams
Part 2 (treatment-naïve patients):The percentage of patients who achieve complete response (CR) | up to 18 weeks
  CR rates at the end of chemotherapy
Part 2 (relapsed or refractory patients):The percentage of patients who achieve complete response (CR) | up to 26 weeks
  CR rates at the end of treatment(including chemotherapy and radiation)
Part 2 (relapsed or refractory patients):The percentage of patients who achieve partial response (PR) | up to 26 weeks
  PR rates at the end of treatment(including chemotherapy and radiation)

SECONDARY OUTCOMES:
Part 1 the preliminary antitumor efficacy: complete response rate (CR) | up to 26 weeks
  the percentage of patients who achieve complete response (CR)（including at the end of chemotherapy and at the end of treatment）
Part 1 the preliminary antitumor efficacy：overall response rate (ORR) | up to 26 weeks
  the percentage of patients who achieve complete response (CR）and partial response (PR)（including at the end of chemotherapy and at the end of treatment）
Part 1 the preliminary antitumor efficacy:disease control rate (DCR) | up to 26 weeks
  the percentage of patients who achieve complete response (CR）、partial response (PR) and stable disease（SD）（including at the end of chemotherapy and at the end of treatment）
Part 1: The pharmacokinetic parameters Cmax | At the end of Cycle 1 and Cycle 3 (each cycle is 21 days)
  maximum concentration(Cmax)
Part 1: The pharmacokinetic parameters AUC0-t | At the end of Cycle 1 and Cycle 3 (each cycle is 21 days)
  area under the curve from zero to the time point（AUC0-t）
Part 2 (treatment-naïve patients):The preliminary antitumor efficacy complete response rate (CR) | up to 26 weeks
  the percentage of patients who achieve complete response (CR)（including at the end of chemotherapy and at the end of treatment）
Part 2 (treatment-naïve patients):The preliminary antitumor efficacy overall response rate (ORR) | up to 26 weeks
  the percentage of patients who achieve complete response (CR）and partial response (PR)（including at the end of chemotherapy and at the end of treatment）
Part 2 (treatment-naïve patients):The preliminary antitumor efficacy disease control rate (DCR) | up to 26 weeks
  the percentage of patients who achieve complete response (CR）、partial response (PR) and stable disease（SD）（including at the end of chemotherapy and at the end of treatment）
Part 2 (treatment-naïve patients):The preliminary safety index | through study completion, an average of 1 year
  The incidence and severity of adverse events (AEs), abnormalities in clinical laboratory assessments, ECGs, vital sign assessments, and physical exams
Part 2 (relapsed or refractory patients): The preliminary antitumor efficacy | up to 26 weeks
  disease control rate (DCR)：the percentage of patients who achieve complete response (CR）、partial response (PR) and stable disease（SD）（including at the end of chemotherapy and at the end of treatment）

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liu, Principal Investigator — 39 Lianhuachi East Road, Haidian Dist., Beijing, China
Locations (1):
- the Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No